CLINICAL TRIAL: NCT07302958
Title: Telerehabilitation, Face-to-Face Exercises, and a Mixed Model in Chronic Non-Specific Neck Pain
Acronym: TR Neck pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ahmad Fallatah, Dr. Amr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR,Face to Face, mix model NP
Record Dates: First submitted 2025-12-08; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: Telerehabilitation; Chronic Non specific Neck pain; Face to face physiotherapy
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real-time Video-Guided Neck Exercises (Tele-rehabilitation) (Experimental): Participants in this arm receive real-time, synchronous tele-rehabilitation sessions delivered via Microsoft Teams video conferencing platform. A licensed physiotherapist provides live supervision, real-time feedback, and technique correction throughout each session. This arm tests the effectiveness of remote delivery of structured neck exercises with synchronous clinician guidance.
  Interventions: Other: Real-Time Video-Guided Neck Exercises (Tele-Rehabilitation)
- In-Person Supervised Neck Exercises (Face-to-Face) (Experimental): Participants in this arm receive traditional, in-person supervised exercise sessions at a clinical facility. A licensed physiotherapist provides hands-on guidance, manual corrections, and real-time feedback during each session. This arm serves as the standard care comparison and tests the effectiveness of conventional face-to-face delivery.
  Interventions: Other: In-Person Supervised Neck Exercises (Face-to-Face)
- Hybrid Tele-rehabilitation and In-Person Exercises (Mixed Model) (Experimental): Participants in this arm receive a novel 50/50 hybrid intervention combining equal proportions of tele-rehabilitation and face-to-face sessions delivered in alternating weekly blocks. Weeks with odd numbers (1, 3, 5) consist of three in-person face-to-face sessions, while weeks with even numbers (2, 4, 6) consist of three tele-rehabilitation sessions. This arm tests whether a hybrid approach optimizes accessibility, adherence, and clinical outcomes by combining the convenience of remote delivery with the benefits of in-person supervision.
  Interventions: Other: Hybrid Tele-Rehabilitation and In-Person Exercises (Mixed Model)

INTERVENTIONS:
Other: Real-Time Video-Guided Neck Exercises (Tele-Rehabilitation) — Intervention 1: Real-Time Video-Guided Neck Exercises (Tele-Rehabilitation)
  How the Intervention is Administered:
  Delivery Method: Real-time video conferencing App
  Frequency: 3 sessions per week
  Duration: 6 weeks (18 total sessions)
  Session Length: 45-60 minutes per session
  Supervision: Live physiotherapist supervision with real-time feedback and exercise modification
  Setting: Participant's home or preferred location with stable internet connection
  Materials Provided:
  Illustrated exercise guide (provided digitally and in print)
  Access to video conferences for sessions
  Optional: Resistance bands for home use
  Arms: Real-time Video-Guided Neck Exercises (Tele-rehabilitation)
Other: In-Person Supervised Neck Exercises (Face-to-Face) — How the Intervention is Administered:
  Delivery Method: In-person supervised sessions at clinical facility
  Frequency: 3 sessions per week
  Duration: 6 weeks (18 total sessions)
  Session Length: 45-60 minutes per session
  Supervision: Direct physiotherapist supervision with hands-on guidance and real-time feedback
  Setting: Clinical rehabilitation facility
  Arms: In-Person Supervised Neck Exercises (Face-to-Face)
Other: Hybrid Tele-Rehabilitation and In-Person Exercises (Mixed Model) — How the Intervention is Administered:
  Delivery Method: Alternating weekly blocks of tele-rehabilitation (video conferencing and face-to-face sessions
  Frequency: 3 sessions per week (alternating delivery)
  Duration: 6 weeks (18 total sessions: 9 tele-rehabilitation + 9 face-to-face)
  Session Length: 45-60 minutes per session
  Supervision: Live physiotherapist supervision for both modalities
  Setting: Mixed (participant's home for tele-rehabilitation weeks; clinical facility for face-to-face weeks)
  Weekly Schedule:
  • Weeks 1, 3, 5: Three face-to-face sessions per week at clinical facility
  • Weeks 2, 4, 6: Three tele-rehabilitation sessions per week via Microsoft Teams
  Materials Provided:
  • Illustrated exercise guide (provided in both digital and print formats)
  • Access to video conferencing App for tele-rehabilitation sessions
  • Access to clinical facility equipment during face-to-face weeks
  • Optional: Resistance bands for home use during tele-rehabilitation week
  Arms: Hybrid Tele-rehabilitation and In-Person Exercises (Mixed Model)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of different physical therapy delivery models in treating chronic non-specific neck pain in adults aged 20-40 years with a history of neck pain for three months or longer.

The main questions it aims to answer are:

* Which approach (tele-rehabilitation, face-to-face exercises, or a mixed model) is most effective at reducing neck pain intensity and functional disability?
* Are there significant differences between the three models in improving cervical range of motion, kinesiophobia (fear of movement), patient satisfaction, and adherence to the exercise program?

Researchers will compare three groups to see if the delivery model affects outcomes:

1. A tele-rehabilitation group receiving real-time, video-guided exercise sessions.
2. A face-to-face group receiving traditional, in-person supervised exercise sessions.
3. A mixed-model group receiving a combination of both tele-rehabilitation and face-to-face sessions.

Participants will:

* Be randomly assigned to one of the three groups.
* Engage in a structured exercise program for 45-60 minutes per session, three times a week for six weeks.
* Follow a phased exercise protocol that begins with mobility and pain reduction, progresses to strengthening, and finishes with endurance and functional training.
* Complete assessments for pain, disability, range of motion, and other outcomes at the beginning and end of the 6-week intervention, with a final follow-up at 3 months.

ELIGIBILITY:
Inclusion Criteria

Patients will be included in the study if they fulfil the following criteria:

* Adults (20-40 years) with chronic non-specific neck pain (≥3 months' duration).
* Participants with stable internet, and experienced in using either computer, laptop, tablet, or smartphone.

Exclusion Criteria

Patients will be excluded if they had:

1. Neck pain due to specific pathologies (e.g., fractures, infections, or malignancies) and severe neurological deficits.
2. History of neck surgery.
3. Participants with cognitive impairments or language barriers that would prevent them from following the interventions.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Disability | • Baseline (Week 0, before intervention begins) • Within 1 week post-treatment (Week 6, immediately after final intervention session) • 3 months post-treatment (Month 3, 12 weeks after completion of intervention)
  The Neck Disability Index is the most widely used and validated instrument for assessing the impact of neck pain on patients' functional activities and disability. The NDI-AR consists of 10 items covering functional domains: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 (no disability) to 5 (complete disability), with a maximum total score of 50.
Neck Pain Intensity | • Baseline (Week 0, before intervention begins) • Within 1 week post-treatment (Week 6, immediately after final intervention session) • 3 months post-treatment (Month 3, 12 weeks after completion of intervention
  The Visual Analogue scale is a self-reported, unidimensional measure of pain intensity. Participants mark their current pain level on a 10-centimeter line, where 0 represents "no pain" and 10 represents "worst pain imaginable.
Range of motion | • Baseline (Week 0, before intervention begins) • Within 1 week post-treatment (Week 6, immediately after final intervention session) • 3 months post-treatment (Month 3, 12 weeks after completion of intervention.
  The CROM device is a non-invasive, objective measurement tool designed specifically for assessing cervical spine mobility. The device measures cervical motion in six planes: flexion, extension, right lateral flexion, left lateral flexion, right rotation, and left rotation. Measurements are recorded in degrees.

SECONDARY OUTCOMES:
Kinesiophobia | • Baseline (Week 0, before intervention begins) • Within 1 week post-treatment (Week 6, immediately after final intervention session) • 3 months post-treatment (Month 3, 12 weeks after completion of intervention)
  The Tampa Scale of Kinesiophobia is a 17-item self-report questionnaire designed to assess the fear of [re]injury associated with physical movement. Respondents rate each item on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("strongly agree"). The total score ranges from 17 to 68, with higher scores indicating greater fear of movement and [re]injury
Patient Satisfaction | • Baseline (Week 0, before intervention begins) • Within 1 week post-treatment (Week 6, immediately after final intervention session)
  The Patient Satisfaction Questionnaire (PSQ-18) is a validated short-form instrument originally developed by the RAND Corporation to measure patient satisfaction with medical care. The PSQ-18 is an 18-item version that retains the essential psychometric qualities of the full-length PSQ-III while providing a practical and comprehensive assessment.
Adherence to Treatment | • Throughout the 6-week intervention period (Weeks 1-6, continuous tracking at each session) • Final adherence rate calculated within 1 week post-treatment (Week 6, at completion of intervention)
  Adherence to treatment is assessed through systematic attendance tracking and session completion records. An attendance sheet is used to register participant attendance at each session with the date and session number. Adherence is calculated as the percentage of completed sessions relative to the total number of prescribed sessions (18 sessions over 6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mohamed Ibrahim, Assistant Professor, Principal Investigator — Cairo University; Moaaz Ragab Riyad, Lecturer of Physical therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennell KL, Nelligan R, Dobson F, Rini C, Keefe F, Kasza J, French S, Bryant C, Dalwood A, Abbott JH, Hinman RS. Effectiveness of an Internet-Delivered Exercise and Pain-Coping Skills Training Intervention for Persons With Chronic Knee Pain: A Randomized Trial. Ann Intern Med. 2017 Apr 4;166(7):453-462. doi: 10.7326/M16-1714. Epub 2017 Feb 21. PMID 28241215
- [Background] Barbosa JC, Comachio J, Marques AP, Saragiotto BT, Magalhaes MO. Effect of a telerehabilitation exercise program versus a digital booklet with self-care for patients with chronic non-specific neck pain: a protocol of a randomized controlled trial assessor-blinded, 3 months follow-up. Trials. 2023 Sep 28;24(1):616. doi: 10.1186/s13063-023-07651-z. PMID 37770963
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Neves Antonio GL, Almeida MQ, Avila MA, de Noronha MA, Approbato Selistre LF. Efficacy of telerehabilitation exercise in patients with chronic neck pain: a protocol for a non-inferiority randomized controlled trial. Pain Manag. 2023 Sep;13(9):497-507. doi: 10.2217/pmt-2023-0070. Epub 2023 Oct 18. PMID 37850374